CLINICAL TRIAL: NCT00829699
Title: Metabolic Causes of Thrombosis in Type 2 Diabetes Mellitus, Question 3
Brief Title: Metabolic Causes of Thrombosis in Type 2 Diabetes Mellitus
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Stephen N. Davis, MBBS, Professor, University of Maryland, Baltimore
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: HP-00044874; RFAHL04016
Record Dates: First submitted 2009-01-23; First posted 2009-01-27 (Estimated); Last update posted 2019-09-12 (Actual); Status verified 2019-09

CONDITIONS: Type 2 Diabetes
Keywords: endothelial function; fibrinolytic balance
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — soybean oil, phospholipid emulsion

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1 (Experimental): Euinsulinemic (low insulin infusion) Euglycemic (normal blood glucose levels) glucose clamp with lipid (fat) infusion
  Interventions: Procedure: euinsulinemic euglycemic glucose clamp
- 2 (Experimental): Euinsulinemic Hyperglycemic (high glucose levels) glucose clamp with lipid infusion
  Interventions: Procedure: euinsulinemic hyperglycemic glucose clamp
- 3 (Experimental): Hyperinsulinemic (High dose insulin) euglycemic glucose clamp with lipid infusion
  Interventions: Procedure: Hyperinsulinemic euglycemic glucose clamp
- 4 (Experimental): Hyperinsulinemic hyperglycemic (high glucose level) glucose clamp with lipid infusion
  Interventions: Procedure: Hyperinsulinemic hyperglycemic glucose clamp

INTERVENTIONS:
Procedure: euinsulinemic euglycemic glucose clamp — euinsulinemic euglycemic glucose clamp with lipid infusion 48 ml/hr for 4 hours
  Other Names: Intralipid
  Arms: 1
Procedure: euinsulinemic hyperglycemic glucose clamp — euinsulinemic hyperglycemic glucose clamp with lipid infusion at 48 ml/hr for 4 hours
  Other Names: Intralipid
  Arms: 2
Procedure: Hyperinsulinemic euglycemic glucose clamp — Hyperinsulinemic euglycemic glucose clamp with lipid infusion at 48 ml/hr for 4 hours
  Other Names: Intralipid
  Arms: 3
Procedure: Hyperinsulinemic hyperglycemic glucose clamp — Hyperinsulinemic hyperglycemic glucose clamp with lipid infusion at 48 ml/hr for 4 hours
  Other Names: Intralipid
  Arms: 4

SUMMARY:
The purpose of this study is to learn more about why patients with diabetes have increased heart attacks, strokes and other illnesses due to blood clots causing blockage of a blood vessel. The proposed protocol will study the separate and combined effects of high glucose and high fats on certain cardiovascular responses in Type 2 DM.

DETAILED DESCRIPTION:
Currently 75-80% of diabetes mellitus (DM) patients die due to thrombotic causes. Data from the Centers for Disease Control and Prevention released in 2000 indicated that mortality due to coronary artery disease is decreasing except in individuals with diabetes. Clearly the disordered metabolism, which includes abnormal metabolism of fats resulting in higher triglyceride and free fatty acid blood levels, occurring in diabetes predisposes these individuals to increased thrombotic events. Unless the underlying mechanisms responsible for these events can be identified, there will be an unprecedented number of diabetic patients suffering thrombotic episodes in the next 10 years.

The specific aims of this study are to determine the effects of elevated free fatty acids and hyperglycemia (high glucose)on endothelial function and thrombolytic balance in patients with type 2 diabetes, and to determine the effects of increased insulin in this setting.

ELIGIBILITY:
Inclusion Criteria

* 16 Type 2 diabetic patients age 18 - 60 yrs
* 16 Non-diabetic controls age 18-60 yrs
* Body mass index >20 kg/m2
* Female volunteers of childbearing potential: negative urine pregnancy test
* Volunteers over 40 years old: an ECG with no clinically significant conduction or ischemic changes.
* For those with type 2 diabetes: HBA1C > 5.5%
* For those with type 2 diabetes: C-peptide >0.2 nmol, If C-peptide is abnormal or there is a clinical suspicion for type 1 diabetes, MODY or LADA, anti-islet cell and anti-GAD antibodies will be assessed to establish the diagnosis of type 2 diabetes vs. type 1/LADA/MODY.
* PT (time) 12.8-14.6 seconds, PTT (time) 25-38 seconds

Exclusion Criteria

* Any current disease condition that alters carbohydrate metabolism (other than type 2 DM) and/or evidence for clinically significant cardiac disease
* Uncontrolled hypertension
* Pregnancy
* Subjects unable to give voluntary informed consent
* Subjects with history of pancreatitis
* Subjects on anticoagulant drugs, anemic, or with known bleeding diseases
* Subjects with history of GI bleeding requiring treatment
* Tobacco Use
* Subjects with history of heparin-induced thrombocytopenia or heparin allergy
* Subjects with severe egg or legume (soybean) allergy
* Abnormal results following screening tests and physical examination that is clinically significant:

Medical history/Physical Exam Exclusion Criteria

* Fever greater than 38 degrees C at screening or study initiation
* Uncontrolled severe hypertension (i.e., blood pressure greater than 160/100)
* Cardiac Abnormalities (e.g. Heart Failure, Arrhythmia, Cardiomyopathy, ischemic tachycardia, S-T segment deviations, etc.,) from history or ECG testing in subjects > 40 years old.
* Diagnosed Pneumonia
* Hepatic Failure/Jaundice
* Clinically significant coagulopathy
* Renal Failure
* Acute Cerebrovascular/ Neurological deficit

Screening Laboratory Tests Exclusion Criteria according to protocol

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2009-07; Primary Completion 2013-06 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Percent change in flow mediated dilation of brachial artery | 4 hours

SECONDARY OUTCOMES:
Change in Lipid measures | 4hours

CONTACTS AND LOCATIONS:
Overall Officials: Stephen N. Davis, MD, Principal Investigator — University of Maryland, Baltimore
Locations (1):
- Univerisity of Maryland, Baltimore, Baltimore, Maryland, United States